CLINICAL TRIAL: NCT04169100
Title: Novel Form of Acquired Long QT Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Narrows Institute for Biomedical Research (Other)
Collaborators: VA New York Harbor Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Deana Lazaro, Chief of Rheumatology, Narrows Institute for Biomedical Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ORD01372
Record Dates: First submitted 2019-11-14; First posted 2019-11-19 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Long QT Syndrome; Connective Tissue Diseases; Rheumatoid Arthritis
Keywords: cytokines
MeSH Terms: conditions — Long QT Syndrome; Connective Tissue Diseases; Arthritis, Rheumatoid | interventions — Prednisone

STUDY DESIGN:
Intervention Model Description: Single group, Preventative care, Proof of concept study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Prednisone Group (Experimental): These patients have CTD and QTc over 500 msec. Prednisone is administered as a preventative measure against arrhythmia via QTc shortening.
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Prednisone — We propose to test whether QT prolongation is reversible with moderate doses of prednisone in patients with QT interval greater than 500 msec.

SUMMARY:
The goal of this study is to determine whether anti-Ro/SSA antibodies are associated with acquired QT prolongation in subjects with connective tissue disease. The investigators will investigate whether gender or race influence correlation between anti-Ro antibody status and prolonged QT interval and the role of inflammatory cytokines in association with anti-Ro antibodies and QT prolongation. The investigators propose to add an additional objective to test whether QT prolongation is reversible with moderate doses of prednisone in patients with QT interval greater than 500 msec.

DETAILED DESCRIPTION:
There are two parts to this study. First, the investigators propose a prospective, observational study of subjects with connective tissue disease (CTD). Data on CTD diagnosis, disease activity, medications, electrolytes, anti-Ro Ab status, QT interval and serum for measurement of inflammatory markers and cytokines will be collected. Please see the research strategy for details of the protocol. The investigators expect that QTc prolongation will have a positive correlation with anti-Ro Ab positivity, elevated measures of inflammatory markers and higher levels of inflammatory cytokines, especially IL-6.

The second part of the study will include a subgroup of subjects who have QTc prolongation of more than 500 milliseconds. This is a proof of concept study to investigate whether immunosuppressive treatment with moderate dose of prednisone will reduce QTc in CTD patients exhibiting an excessive QTc prolongation of >500msec. Patients enrolled in the prospective observational study with QTc prolongation of more than 500 msec will receive oral prednisone 40mg daily for 3 days followed by 20mg for eleven days (a total of 2 weeks) with the goal to shorten or normalize the prolonged QTc. Other factors that may cause prolonged QTc will be evaluated and corrected as needed. Inflammatory markers, cytokines, and QTc will be measured at baseline and serially at days 3 and 14 (end of treatment). The investigators will monitor changes in QTc during three 24-hour periods during treatment at baseline, day 3 and day 14. Risks of prednisone include elevated serum glucose levels, edema, increased risk of infection and blood pressure elevation. The dosage and duration of prednisone used in this study is similar to that given for a severe allergic reaction. The PI will monitor the patients for potential side effects which will immediately be addressed.

ELIGIBILITY:
Inclusion Criteria:

- Patients enrolled in New York Harbor Healthcare System with connective tissue disease

Exclusion Criteria:

* Atrial fibrillation
* Intraventricular conduction delay with wide QRS complex
* Acute medical conditions
* Drug overdose
* Hypothermia
* Known diagnosis or family history of hereditary Long QT syndrome, complete bundle brunch block, ventricular paced rhythm, profound bradycardia and tachycardia, and uncorrected hypothyroidism

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2011-09-28 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Corrected QT Interval | Baseline and at 14 days
  QT interval to be measured on electrocardiogram

SECONDARY OUTCOMES:
Change in Cytokine Levels | Baseline and at 14 days
  IL-1β, sTNFR1, TNFα, IL-10, IL-6, and α-interferon
Change in ESR | Baseline and at 14 days
  Inflammatory Marker
Change in CRP | Baseline and at 14 days
  Inflammatory Marker

CONTACTS AND LOCATIONS:
Locations (1):
- VA New York Harbor Healthcare System, NY and Brooklyn Campuses, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified can be shared upon request. We do not anticipate the generation or development of any model organism or unique reagent from this study. If any new model organism or reagent is generated then we will make them available to other researchers upon request via the VA New York Harbor Healthcare System Technology Transfer office.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available from the time of publication and will be kept for a minimum of 5 years.
Access Criteria: Data will be shared upon written request to the principal investigator.